CLINICAL TRIAL: NCT02190617
Title: Guidelines to Practice: Reducing Asthma Health Disparities Through Guideline Implementation
Acronym: G2P
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Public Health - Seattle and King County (Other Government)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None
Other Study IDs: AS1307-05498
Record Dates: First submitted 2014-07-11; First posted 2014-07-15 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2014-07

CONDITIONS: Asthma
Keywords: Asthma; Guidelines; Community Health Worker
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Enhanced Clinic+ Unified Management Plan (Active Comparator): Patients in study arm will receive:
  * Enhanced Clinic Intervention
  * Enhanced Health Plan
  * Unified Management Plan
  Interventions: Behavioral: Enhanced Clinic+ Unified Management Plan
- CHW Home Visit Only (Active Comparator): Patients in study arm will receive:
  * CHW Home Visit
  * Usual clinic care with enhanced health plan
  Interventions: Behavioral: CHW Home Visit Only
- Enhanced Clinic+ Unified Plan+ CHW (Active Comparator): Patients in study arm will receive:
  * CHW Home Visit
  * Enhanced Clinic intervention
  * Enhanced health plan
  * Unified asthma management plan
  Interventions: Behavioral: Enhanced Clinic+ Unified Plan + CHW
- Usual Care (No Intervention): -Usual clinic care with enhanced healthplan

INTERVENTIONS:
Behavioral: Enhanced Clinic+ Unified Plan + CHW — * Unified asthma management plan and asthma support team coordination: A support team will partner with each patient to develop a single asthma management plan. An EMR will provide a web-based platform for sharing the unified asthma management plan.
  * Home visit intervention: Community health workers will provide in-home tailored asthma support and conduct follow-up to support patient actions to improve asthma control based on unified asthma management plan.
  * Enhanced clinic intervention: Intervention clinics will implement a multicomponent intervention that will include decision support, audit and feedback, provider and staff education, asthma champions, team-based care, and spirometry, all supported by EMR enhancements and clinic systems redesign.
  Other Names: -Enhanced Clinic; -CHW Home Visits; -Unified Management plan
  Arms: Enhanced Clinic+ Unified Plan+ CHW
Behavioral: Enhanced Clinic+ Unified Management Plan — * Unified asthma management plan and asthma support team coordination: A support team (clinicians, CHWs and plan care managers) will partner with each patient to develop a single asthma management plan. An EMR will provide a web-based platform for sharing the unified asthma management plan and enhancing communications among care team.
  * Enhanced clinic intervention: Intervention clinics will implement a multicomponent intervention that will include decision support, audit and feedback, provider and staff education, asthma champions, team-based care, and spirometry, all supported by EMR enhancements and clinic systems redesign.
  Other Names: -Unified Management Plan; -Enhanced Clinic Intervention
  Arms: Enhanced Clinic+ Unified Management Plan
Behavioral: CHW Home Visit Only — -Home visit intervention: Community health workers will provide in-home tailored asthma support: assess asthma self-management knowledge and skills, conduct a home environmental assessment focused on asthma triggers, and conduct follow-up visits to support patient actions to improve asthma control based on unified asthma management plan.
  Other Names: -CHW Home Visit Intervention
  Arms: CHW Home Visit Only

SUMMARY:
The primary hypothesis the investigators will test is that that improving asthma guideline implementation and providing patients with a unified asthma management plan using a multi-component and multilevel intervention will improve patient-centered asthma outcomes compared to health plan case management, passive guideline dissemination and provider education.

DETAILED DESCRIPTION:
The study will use a factorial randomized controlled design to assess the comparative effectiveness of the following interventions among 8 community health centers and 550 patients with:

* Health plan enhanced intervention plus traditional provider education: Health plans will enhance case management support, monitor medication fills, and increase passive guideline dissemination. Traditional provider education will consist of implementation of the PACE asthma education program. Note that all participants and clinics will receive this intervention. In effect, this will be the base active comparator arm of the study.
* Home visit intervention: Community health workers will provide in-home tailored asthma support: assess asthma self-management knowledge and skills, conduct a home environmental assessment focused on asthma triggers, and conduct follow-up visits to support patient actions to improve asthma control based on unified asthma management plan.
* Enhanced clinic intervention with system integration: Clinics will implement a multi-component intervention that includes decision support, audit and feedback, provider and staff education, team-based care, and training and feedback in implementing office spirometry and allergy testing. EHR enhancements and clinic systems redesign will support this work. The EHR will also provide a platform for sharing a common asthma management plan and enhancing communications among care team members (clinicians, CHWs, plan case managers).

All four intervention groups will receive enhanced health plan intervention + provider education. The four study arms will receive the following additional different interventions: (a) usual clinic care; (b) a + home visit, (c) enhanced clinic care + system integration, and (d) c + home visit.

ELIGIBILITY:
Inclusion Criteria:

* Age 5-75
* Provider-verified diagnosis of asthma
* Have uncontrolled asthma
* Primary language of English,Spanish or Vietnamese
* Patient of Neighborcare or HealthPoint Health
* Insured by Molina Healthcare or Community Health Plan of Washington

Exclusion Criteria:

* Patient planning to leave Neighborcare or Healthpoint Health within the next 12 months
* Household appearing to be unsafe for a visit by a community health worker
* Co-existing medical conditions that make asthma control a low priority for patient management or that confound outcome measurement or that preclude participation in self-management
* Participation in another asthma research study

Ages: 5 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 550 (Estimated)
Dates: Start 2014-12; Primary Completion 2016-10 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Symptom free days | 12 Months
  Measured by questionnaire: Days without cough, wheeze, chest tightness, shortness of breath, nocturnal wakening from symptoms or activity limitation due to asthma in past 2 weeks.
Asthma control | 12 Months
  Measured by questionnaire and spirometry. Asthma Control Adults: Asthma Control Test and EPR3 categories Asthma Control Children: cACT and EPR3 categories
Asthma-related Quality of Life | 12 Months
  Measured by questionnaire.
  Adults:
  * Mini Asthma Quality of Life Questionnaire
  Children 7-17:
  * Pediatric Asthma Quality of Life Questionnaire
  Children 5-6:
  * Pediatric Asthma Caregiver Quality of Life Scale

SECONDARY OUTCOMES:
Nocturnal wakening | 12 Months
  Measured by questionnaire: Nights wakened in the past two weeks due to asthma.
Asthma exacerbations | 12 Months
  Measured by questionnaire: Need for oral steroids (3+ day course), hospitalization, ED visit or unscheduled clinic visit for worsening asthma in past 12 months
Pulmonary function | 12 Months
  Measured by spirometry: Post-bronchodilator FEV1 and FEV1 /FVC and change in pre-post bronchodilator FEV1 and FEV1 /FVC182 using EasyOne Diagnostic spirometer
FeNO (Fractional exhaled Nitric Oxide) | 12 Months
  Measured by portable handheld device: Online measurement of ppb in exhaled breath at 50 L/s (<25 ppb indicates normal value.)
Beta-agonist use | 12 Months
  Measured by questionnaire and claims data: Days using Beta-agonist medication in past 2 weeks
Oral steroid use | 12 Months
  Measured by questionnaire and claims data: Courses of steroids (3+ day course) in past 12 months
Controller use | 12 Months
  Measured by claims data: Controller to total asthma medication ratio > 0.5
Asthma-related urgent health services utilization | 12 Month
  Measured by questionnaire and administrative data: Urgent clinic visits, emergency department visits, and hospitalizations during past three months and past year
Missed work or school days | 12 Months
  Measured by questionnaire: Number of school or work days missed in past two weeks.
General Health Status | 12 Months
  Measured by questionnaire:
  Adults: SF-12 Health Survey Children: SF -10 Health Survey

CONTACTS AND LOCATIONS:
Overall Officials: James Stout, MD, Principal Investigator — University of Washington
Locations (1):
- Public Health -- Seattle & King County, Seattle, Washington, United States